CLINICAL TRIAL: NCT06920238
Title: A Phase I Single-Arm Trial to Test the Use of a Generative AI (Gen-AI) Chatbot for Anxiety and Depression Among Persons With Cannabis Use Disorder (CUD)
Brief Title: Use of a Generative AI (Gen-AI) Chatbot for Anxiety and Depression Among Persons With Cannabis Use
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Trustees of Dartmouth College (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Nicholas Jacobson, Associate Professor, Trustees of Dartmouth College
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: STUDY00033219; 5P30DA029926-14 (NIH)
Record Dates: First submitted 2025-03-10; First posted 2025-04-09 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Cannabis Use Disorder; Anxiety; Depression, Anxiety; Depression - Major Depressive Disorder
Keywords: Artifical Intelligence; Generative AI; Generative Artificial Intelligence; Therabot; Therabot-CALM; Cannabis Use Disorder; Anxiety; Depression; Chatbot; Cannabis Use; Drug Abuse; Drug Use; Drug Use Disorder; Interview; Screening; Application; REDCap; post-intervention measures; System Usability Scale; Treatment Acceptability and Adherence Scale; Cannabis Use Disorders Identification Test - Revised; Cannabis Use Disorders Identification Test; Quantity of Cannabis Use Inventory; Patient Health Questionnaire for depression; generalized anxiety disorder screener; DSM-5; Zoom
MeSH Terms: conditions — Anxiety Disorders; Depression; Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: Therabot-CALM Model
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Therabot-CALM (Experimental): Participants will engage in three one-hour interviews and a 4-week clinical trial where they may interact with Therabot-CALM as much or as little as they want.
  Interventions: Device: Therabot-CALM

INTERVENTIONS:
Device: Therabot-CALM — Therabot is a generative-AI-driven mobile app designed to provide mental health treatment. The feasibility of Therabot-CALM, an adapted Therabot application, is being tested for the future use of treating co-occurring substance use disorders and anxiety and/or depression. The primary purpose of this study is application feasibility.

SUMMARY:
The goal of this clinical trial is to learn if Therabot-CALM (Cannabis, Anxiety, Low Mood) has acceptability among users and could work to improve the symptoms of persons with cannabis use disorder and anxiety and/or depression. The main question it aims to answer is:

What is the usability, feasibility, and acceptability of Therabot-CALM in persons with Cannabis Use Disorder and Anxiety and/or Depression?

Participants will

* Take a screening questionnaire
* Participate in two virtual 1-hour interviews to provide feedback on app design and suggest features.
* Engage with Therabot-CALM in a 4-week clinical trial and provide feedback on their app experience in a third virtual interview

DETAILED DESCRIPTION:
Participants will complete a two-stage screening process via REDCap to determine their eligibility for enrollment. Participants who meet criteria and provide informed consent will be enrolled and participate in three interviews and the 4-week clinical trial.

After the first interview, researchers will fine-tune Therabot-CALM based on feedback received during the interview. After the second interview, experts by experience (EBEs) will engage with Therabot-CALM at least once per day for 4 weeks. After the clinical trial period, participants will receive an email with a link to complete the post-intervention measures delivered via REDCap, including the System Usability Scale (SUS), Treatment Acceptability and Adherence Scale (TAAS), Cannabis Use Disorders Identification Test - Revised (CUDIT-R), the Daily Sessions, Frequency, Age of Onset, and Quantity of Cannabis Use Inventory (DFAQ-CU), the 9-item Patient Health Questionnaire for depression (PHQ-9), and the 7-item generalized anxiety disorder screener for DSM-5 (GAD-7). Participants will then be asked to return for a third interview to provide feedback on their experience with Therabot-CALM.

Researchers will use the IDEAS (Innovate, Develop, Evaluate, Adapt, Scale) Impact Framework to plan and conduct three, one-on-one interviews with a trained research assistant (RA). Each interview script will be developed using the IDEAS Impact Framework and follow a semi-structured design, such that the RA will follow a set of questions, with as-needed probing for follow-up. Interviews will be recorded via a virtual platform.

ELIGIBILITY:
Inclusion Criteria:

* Is 18 years or older.
* Meet criteria for current CUD (CUDIT-R>=12) and MDD (PHQ-9>=10), and/or GAD (GAD-7>=10).
* Have reliable access to the internet and a compatible device for Therabot-CALM.
* Have willingness and capacity to provide informed consent and commit to participating in all assessments and interventions during the study.
* Attend the first interview.

Exclusion Criteria:

* Moderate to High risk of STBs as determined by the C-SSRS or baseline questionnaires.
* Current psychosis (as determined by brief psychosis screen).
* Current participation in another digital mental health intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-04-13 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Feasibility | From enrollment to the end of the third interview at around 10 months
  Feasibility of the application is measured by engagement rates of participants. Engagement rates will be quantified based on the frequency and duration of interactions with the application during the clinical trial period.
Usability | From enrollment to the end of the third interview at around 10 months
  Usability is measured by participant responses on the System Usability Scale (SUS). The SUS score will range from 0 to 100, where higher scores indicate better usability.
Acceptability | From enrollment to the end of the third interview at around 10 months
  Acceptability is measured by the Treatment Acceptability and Adherence Scale (TAAS), the Likert-style satisfaction rating scale to assess satisfaction with Therabot-CALM. The TAAS scale will range from 0 to 100, where higher scores indicate higher acceptability. The Likert-style satisfaction rating scale will range from 1 to 5, with 1 indicating very dissatisfied and 5 indicating very satisfied.

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas C Jacobson, Ph.D., Principal Investigator — Center for Technology and Behavioral Health, Geisel School of Medicine, Dartmouth College
Locations (1):
- 46 Centerra Parkway, Suite 300, Office #333S, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Heinz, M. V., Mackin, D., Trudeau, B., Bhattacharya, S., Wang, Y., Banta, H. A., Jewett, A. D., Salzhauer, A., Griffin, T., & Jacobson, N. C. (2024). Evaluating Therabot: A Randomized Control Trial Investigating the Feasibility and Effectiveness of a Generative AI Therapy Chatbot for Depression, Anxiety, and Eating Disorder Symptom Treatment. OSF. https://doi.org/10.31234/osf.io/pjqmr
- [Background] Collins AC, Bhattacharya S, Oh JY, Salzhauer A, Taylor CT, Wolitzky-Taylor K, Aupperle RL, Budney AJ, Jacobson NC. Inclusion of Individuals With Lived Experiences in the Development of a Digital Intervention for Co-Occurring Depression and Cannabis Use: Mixed Methods Investigation. JMIR Form Res. 2024 Oct 7;8:e54751. doi: 10.2196/54751. PMID 39374076